CLINICAL TRIAL: NCT03945682
Title: The ASsessment and Physiotherapy managEment of Ataxia in Children Following Surgical Resection of Posterior Fossa Tumour (ASPECT)
Brief Title: The ASsessment and Physiotherapy managEment of Ataxia in Children Following Surgical Resection of Posterior Fossa Tumour
Acronym: ASPECT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alder Hey Children's NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 227917
Record Dates: First submitted 2019-05-08; First posted 2019-05-10 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Ataxia; Posterior Fossa Tumor
Keywords: physiotherapy; surgical resection
MeSH Terms: conditions — Ataxia; Infratentorial Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants will be randomised to one of 2 groups 1. Intervention arm 2. Usual standard of care.
Masking Description: No study drug as part of this RCT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapist (Experimental): Intervention therapist at 2 centres providing 8 week intervention programme 50% embedded qualitative study
  Interventions: Other: Therapist
- Usual Standard of Care (No Intervention): Participants continue with usual care and existing therapy recorded in study diary

INTERVENTIONS:
Other: Therapist — Intervention therapist at 2 centres providing 8 week intervention programme 50% embedded qualitative study
  Arms: Therapist

SUMMARY:
The overall aim of the study is to determine the feasibility of conducting a randomised controlled trial (RCT) studying the effectiveness of physiotherapy intervention (virtual training) in children with ataxia following surgical resection of posterior fossa tumour

DETAILED DESCRIPTION:
Brain tumours are the most common group of solid tumours in children accounting for nearly a quarter of all childhood cancers. There are approximately 500 new cases of central nervous system (CNS) tumours in children/adolescents reported in the UK per year. Although prognosis has improved over the last 30 years, brain tumours remain the leading cause of tumour-associated death in children. Surgical resection is a mainstay of management of children with brain tumours, as for several tumour types there is strong evidence that survival and progression free survival are influenced by the degree of resection. Therefore extensive tumour removal is an operative goal, but the morbidity of surgery along with any subsequent oncological treatment should also be considered. The NICE guidelines for improving outcomes in children and young people with cancer identify that 'Survivors of CNS malignancy are among the neediest of all cancer survivors, because of the effects of the tumour and multimodality therapy, all of which affect neurological, psychological, endocrine and academic function and become more evident with increasing age'.

Children with posterior fossa tumours (PFT), which account for approximately 50% of all childhood brain tumours, have a distinctive set of issues e.g. potential for gross change pre/post operatively, rapid onset of ataxia, hydrocephalus and increased intra-cranial pressure adding deficits distinct from ataxia, in addition to potential problems from any subsequent oncological management such as radiotherapy. Of these issues, ataxia is the predominant motor problem in children with posterior fossa tumours. Ataxia can describe a related number of impairments including upper limb control, balance, gait difficulties, eye movement issues and speech problems. It is a presenting sign in 58-90% of children with posterior fossa tumours. Ataxia and balance problems also persist long term following surgery, Piscione et al found 70% of children with posterior fossa tumours will have long term post-operative balance problems. Lannering et al specified that truncal ataxia was the most disabling motor impairment in children with brain tumours.

Access to neuro-rehabilitation is recognized as crucial in paediatric neuro-oncology with physiotherapy integral to this; yet there is no consensus as to the type, intensity or timing of interventions. A literature review of physical therapy/physiotherapy for children with ataxia (of any origin) was carried out in preparation for this project to confirm the literature gap, and consider interventions that have been of value in other pathologies causing ataxia. Ten papers in total were identified which included three review papers that covered adult and paediatric literature though the data were not separated in the studies to enable consideration of paediatrics as a distinct group. Overall the reviews concurred there was a suggestion of the benefit of physiotherapy (including treadmill training, rehabilitation, virtual training) though treatment modalities were often not consistently defined and evidence was typically of low quality (level III/IV). The recommendations from these reviews are that the next step would be to undertake RCTs (randomised controlled trials) in more homogenous patient groups. Looking at the paediatric literature, there were three case studies identified (and one case series with a population of three adolescents) again in differing diagnoses though none were examining children with brain tumours that is the most common acute cause for ataxia in the paediatric population. The largest paediatric study (n=10) identified through the literature review was a cohort study by Ilg et al evaluating the effect of virtual training. Virtual training refers to the use of computer technologies that provide an interactive environment that requires limb movement to react to on screen game play. Ilgs study found positive results and proposed that virtual training should then complement/supplement therapy treatment tailored according to the individual and continued in the home environment. Virtual training has also been explored in other paediatric populations e.g. cerebral palsy.

Overall the literature review highlighted that there is a gap in the literature regarding physiotherapy intervention for children with ataxia, in particular there is no literature on effectiveness of physiotherapy for children with brain tumours. However, there is an emerging evidence base in adults with ataxia and to a lesser extent paediatric populations as described above, from similar (though non acute) lesions in the cerebellum reporting the benefits of balance therapies including virtual training. This suggests the potential for recovery from ataxia in similar conditions i.e. children with damage to the cerebellum following surgical resection of posterior fossa tumour.

ELIGIBILITY:
Inclusion Criteria:

* Child or young person (4-<18 years) demonstrating ataxia. (For this study, ataxia is currently defined as SARA greater than 2. This definition is taken from data from the CARS study to date, from the cut off threshold value distinguishing no ataxia from mild ataxia)
* 12 months to 3 years following surgical resection of posterior fossa tumour. (This time frame has been selected as this covers the time when the children will typically have completed any adjunct oncology treatment and therefore more emphasis is dedicated to rehabilitation).

Exclusion Criteria:

* Medically unstable/currently undergoing adjunctive treatment e.g. radiotherapy or chemotherapy
* Less than 4 years of age (due to inability to complete standardized assessments)
* Aged 18 or over
* Unable to stand independently for less than one minute or SARA gait item score over 4, either of which would inhibit capacity to complete the training session.
* Presence of co-morbities with the potential to affect the safety of training, such as congenital or acquired disorders causing high risk of falls or lack of comprehension of training tasks, or current musculoskeletal impairments (such as a non-union fracture or fracture currently healing limiting weight-bearing)

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-03-05 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Process Measures | 32 months
  Number of patients identified who meet the inclusion criteria and are then subsequently recruited will be recorded.
Intervention Process Measures | 32 months
  Number of patients who complete all sessions of the intervention will be recorded and the patient's adherence to treatment in the home setting will be noted.

SECONDARY OUTCOMES:
SARA | 32 months
  Scale for the Assessment and Rating of Ataxia
BARS | 32 months
  Brief Ataxia Rating Scale
9HPT | 32 months
  Nine hole peg test
PEDI | 32 months
  Paediatric Evaluation of Disability Index
PedsQL | 32 months
  Brain Tumour Module
BBS | 32 months
  Berg Balance Scale
INAS | 32 months
  Inventory of Non Ataxia Signs. Assessment of compliance (diary)
Subjective Impact | 32 months
  Subjective Impact Likert Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Alder Hey Children's NHS Foundation Trust, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: No